CLINICAL TRIAL: NCT07177157
Title: The Prospective Improved Vitamin D Study for IBD Patients Part 2 (The PIVD Study Part 2)
Brief Title: The Prospective Improved Vitamin D Study for Inflammatory Bowel Disease Patients
Acronym: PIVD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Terry Ponich (Other)
Responsible Party: Sponsor-Investigator, Terry Ponich, Gastroenterology Team Clinician - Victoria Hospital (LHSC), London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WREM: 125544
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis (UC); IBD (Inflammatory Bowel Disease); Crohn Disease (CD)
Keywords: vitamin D; Inflammatory Bowel Disease; IBD; Ulcerative Colitis; Bone Health; Immune Modulation; Crohn Disease (CD)
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Crohn Disease | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D (Experimental): Participants who have IBD (UC or CD) will receive Vitamin D3 and will take a 2000 IU pill daily for 12 months.
  Interventions: Dietary Supplement: Vitamin D3 (Cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (Cholecalciferol) — 2000 IU of Vitamin D daily (1 pill)

SUMMARY:
The aim of this clinical trial is to gain a better understanding of the effect of Vitamin D supplementation on disease activity and overall health. The main questions it aims to answer are:

1. What proportion of IBD patients adhere to Vitamin D supplement recommendations over a 12-month period?
2. Is the ASK-12 Questionnaire valid in measuring adherence among IBD patients?
3. Does the severity of a patient's Crohn's disease effect overall adherence, over a 12-month period?
4. Does the severity of a patient's Ulcerative Colitis disease effect overall adherence, over a 12-month period?
5. Does Vitamin D supplementation affect the health-related Quality of Life for IBD patients?
6. Is 2,000 IU/Day an effective dose to sustain appropriate blood Vitamin D levels among previously Vitamin deficient IBD patients?

Participants will:

* Take 2000 IU of Vitamin D every day for the next 12 months
* Complete 2 surveys, bloodwork and a fecal calprotectin test at the initial, visit, 6 month follow up and 12 month follow up

DETAILED DESCRIPTION:
Upon investigating the literature, despite there being a lot of medication compliance research, there was not much research catered to IBD patient medication management specifically.

Vitamin D supplementation based on immune-modulatory effects alongside its beneficial effects on bone health can lead to reduced rates of osteopenia and osteoporosis in the IBD population. In the treatment of IBD, the major patient care objectives to relieve symptoms and reduce inflammation doesn't leave much time or consideration for other aspects of patient care such as Vitamin D supplementation.

This study will investigate the gastroenterology department at LHSC to assess the current state of adherence and monitoring of Vitamin D and other medications for both Crohn's disease and ulcerative colitis patients. This will be done through a prospective cohort study of patients whose records have stated that they are not currently on Vitamin D. Through assessing overall adherence, foundational understanding of the IBD population will be obtained and the use the ASK-12 questionnaire will be validated. Once done, this would allow for a broader understanding of the patient specific factors affecting individual adherence and lay the foundation for research into ways at increasing adherence among non-adherent individuals.

The overall objective of this study is to estimate the proportion of patients that adhere to Vitamin D supplements. It is the hope that through investigations Vitamin D monitoring and adherence can be standardized at LHSC and long term osteoporosis and osteopenia complications commonly experienced by the IBD patient population can be prevented.

The central hypothesis is that Vitamin D adherence among IBD patients is low and that it is closely related to the patient's IBD disease severity. It is anticipated for this Vitamin D trend to be reversed, as patients may want to stabilize the disease condition and limit acute exacerbations prior to restarting maintenance therapy in the form of Vitamin D treatment.

A clinician as part of the gastroenterology team at Victoria Hospital or St. Joseph's Hospital (Dr. Ponich and other members of VH GI team) who is the primary healthcare contact for the recruited patient will make initial contact with potential participants. Dr. Ponich or another member of the VH GI team will approach the patient in clinic after their visit and ask a member of the research team to discuss the purpose and procedure of the study. The research team member will have the patients fill out a short-written consent form that meets the standards at LHSCRI as submitted in the WREM application. The research team member will obtain written consent from the patient.

Recruited patient's will be provided Vitamin D supplementation and be asked to take 2,000 IU/day. No additional reinforcement will be provided to these patients. At both 6- and 12-month intervals, remaining supplements will be collected, and overall adherence will be assessed. Participants will be asked to complete the EQ-5D-5L to assess their health-related quality of life and the ASK-12 Questionnaire, which will be compared to the pill counts, to determine the validity of ASK-12 among IBD patients. The Patients' IBD will be assessed by performing either a Partial Mayo or CDAI Score as well as completing a fecal calprotectin test. Additionally, participant serum Vitamin D levels will be collected to determine whether adherence to medication resulted in an identifiable increase.

ELIGIBILITY:
Inclusion Criteria:

1. Adults Aged 18-85
2. Diagnosis of IBD (Ulcerative Colitis or Crohn's Disease) within the patient's records based on standard clinical, endoscopic, and radiologic criteria.
3. Patients within outpatient gastroenterology clinics at Victoria Hospital and St. Joseph's Hospital with follow-up appointments within the next 2 years (ongoing IBD care).
4. Participants must have the ability to read, comprehend, and voluntarily provide informed consent without assistance.

Exclusion Criteria:

1. Those who do not meet the inclusion criteria.
2. Those with any concurrent diagnosis of disease that may affect calcium or Vitamin D metabolism (i.e., rheumatoid arthritis or other inflammatory joint disease, thyroid disease, parathyroid disease, primary bone disease, granulomatous disease, sarcoidosis, lymphoma).
3. Those with either renal dysfunction (serum creatinine >0.150 mmol/L) or receiving dialysis were excluded, patients with chronic liver disease, and hypercalcemia (>2.65mmol/L).
4. Those using oral corticosteroids for the management of any disease other than IBD.
5. Those with a history of Vitamin D or calcium supplementation within 6 months prior to the trial.
6. Those who were seen once by the gastroenterology team but never followed up (no ongoing IBD care).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | Enrollment to 12 month follow up
  Assessing the proportion of IBD patients, at both 6 and 12 months, who are adherent to Vitamin D supplementation using pill-counting of supplements provided to them.

SECONDARY OUTCOMES:
Validity of ASK-12 Survey | Enrollment until 12 month follow up
  Determining the validity of the ASK-12 survey, a 12-item Short Health Survey adherence tool will be used to assess adherence rates, among the IBD patients. The ASK-12 Questionnaire detects patient specific barriers to medication adherence, with scores ranging from 12-60 (higher scores indicating a greater non-adherence). The ASK-12 also contains 3 separate subscales: (1) Adherence Behaviors, (2) Health Beliefs, (3) Inconvenience/Forgetfulness.
Quality of Life Assessment | Enrollment until 12 month follow up
  Assessing the change in quality-of-life among IBD patient's using the EQ-5D-5L survey to assess the general health among the patient population. The EQ-5D-5L Health Survey is a 5- item survey that assesses both physical and mental health. There are 5 subcategories that consist of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. There is also a scale where the patient assesses their current overall health ranging from 0 (the worst health they can imagine) to 100 (the best health they can imagine). This tool will be used to compare any changes in health-related quality of life among IBD patients based on their individual rates to supplementations.
Crohn's Disease - Disease Severity | Enrollment until 12 -month follow up
  Assessing the patient's Crohn's Disease severity using the Crohn's disease activity index (CDAI) respectively. The CDAI is a validated tool in assessing disease severity among Crohn's disease patients, with a score >150 indicative of active disease. Any other scores would indicate that the disease is in remission. It will also be looked at by testing fecal calprotectin levels which will allow for comparison of the level of inflammation.
Ulcerative Colitis - Disease Severity | Enrollment until 12-month follow up
  Assessing the patient's Ulcerative Colitis disease severity using the Mayo Disease Activity Index (DAI) respectively. The DAI is a validated tool used in assessing disease severity among Ulcerative Colitis patients, with a score >2 indicative of active disease. Any other scores would indicate that the disease is in remission. It will also be looked at by testing fecal calprotectin levels which will allow for comparison of the level of inflammation.
Impact on Serum Vitamin D Levels | Enrollment until 12 month follow up
  Assessing the effect that providing 2,000 IU/Day of Vitamin D supplements would have on the Serum Vitamin D of IBD patients. Serum Vitamin D levels will be collected and compared to the patient's individual adherence levels using the pill-counting method.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Ponich, MD, Principal Investigator — Victoria Hospital - London Health Sciences Centre
Locations (1):
- Victoria Hospital - London Health Sciences Centre, London, Ontario, Canada